CLINICAL TRIAL: NCT04196192
Title: Febrile Infants - Diagnostic Assessment and Outcome
Acronym: FIDO
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Bristol Royal Hospital for Children (Other); University Hospitals, Leicester (Other); Barts & The London NHS Trust (Other); Children's Health Ireland (Other Government); Royal Hospital for Children Glasgow (Unknown); Royal Belfast Hospital for Sick Children (Unknown)
Responsible Party: Principal Investigator, Thomas Waterfield, Doctor, Belfast Health and Social Care Trust
Other Study IDs: QIP10/12/19HJ
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Meningitis, Bacterial; Bacterial Infections; Urinary Tract Infections
MeSH Terms: conditions — Meningitis, Bacterial; Bacterial Infections; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All infants aged 0-90 days (inclusive) undergoing routine assessments for fever without source.

SUMMARY:
The purpose of this study is to assess how clinicians apply guidance in the assessment of febrile infants presenting the the Emergency Department. The measurable outcomes are:

Primary Objective Report the rates of serious and invasive bacterial infections in febrile infants

Secondary Objectives Report on the predictive value of different clinical features for predicting bacterial infections.

Report on the value of biomarkers for predicting serious and invasive bacterial infections.

Assess the performance of clinical practice guidelines for the assessment of febrile infants.

DETAILED DESCRIPTION:
The assessment of febrile infants is difficult. In the UK and Ireland current guidance advocates that most children under 3 months of age with a fever undergo a full septic screen including lumbar puncture and receive parenteral antibiotics. Approaches in the United States and Europe including the PECARN and StepByStep approach allow for the discharge home of some low risk young infants.

We intend to assess the current approach to febrile infants and compare that to the available clinical practice guidelines. We also intend to determine which clinical and/or laboratory features are most predictive of serious bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Any infant aged 0 to 90 days (inclusive) with a fever of 38 degrees centigrade or higher recorded in the Emergency Department.

Max Age: 90 Days | Sex: All
Age Groups: Child
Study Population: Infants aged 0-90 days (inclusive) with a fever of 38 degrees centigrade or higher recorded in the Emergency Department between the 31/08/2018 and the 01/09/2019.
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Invasive bacterial infection | seven days
  Invasive Bacterial Infection (non-contaminant) confirmed by culture or molecular diagnostic testing of a sterile site i.e. blood or cerebrospinal fluid (CSF). Staphylococcus epidermidis, Propionibacterium acnes, Streptococcus viridans, or Diphtheroides were considered contaminants.
Serious bacterial infections | seven days
  Urinary tract infections defined as growth of ≥100 000 cfu/mL

CONTACTS AND LOCATIONS:
Locations (6):
- Children's Health Ireland, Dublin, Ireland
- United Kingdom (5):
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Bristol Royal Children's Hospital, Bristol
  - Royal Hospital for Children Glasgow, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised datasets not containing any personal data will be available after publication

REFERENCES:
- [Derived] Waterfield T, Foster S, Platt R, Barrett MJ, Durnin S, Maney JA, Roland D, McFetridge L, Mitchell H, Umana E, Lyttle MD; Paediatric Emergency Research in the UK and Ireland (PERUKI). Diagnostic test accuracy of dipstick urinalysis for diagnosing urinary tract infection in febrile infants attending the emergency department. Arch Dis Child. 2022 Dec;107(12):1095-1099. doi: 10.1136/archdischild-2022-324300. Epub 2022 Aug 24. PMID 36002228
- [Derived] Waterfield T, Lyttle MD, Munday C, Foster S, McNulty M, Platt R, Barrett M, Rogers E, Durnin S, Jameel N, Maney JA, McGinn C, McFetridge L, Mitchell H, Puthucode D, Roland D; Paediatric Emergency Research in the UK and Ireland (PERUKI). Validating clinical practice guidelines for the management of febrile infants presenting to the emergency department in the UK and Ireland. Arch Dis Child. 2022 Apr;107(4):329-334. doi: 10.1136/archdischild-2021-322586. Epub 2021 Sep 16. PMID 34531196